CLINICAL TRIAL: NCT01472016
Title: A Multi-Center, Phase 1/1b, Open-Label, Dose Escalation Study of ABT-700, a Monoclonal Antibody in Subjects With Advanced Solid Tumors
Brief Title: Study of ABT-700 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-375
Record Dates: First submitted 2011-10-14; First posted 2011-11-16 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-06

CONDITIONS: Advanced Solid Tumors
Keywords: c-Met overexpression; MET amplification; Neoplasms; h224G11
MeSH Terms: conditions — Neoplasms | interventions — telisotuzumab vedotin; Docetaxel; IFL protocol; Cetuximab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort A (Experimental): ABT-700 will be administered by intravenous infusion at escalating dose levels in 21-day dosing cycles. Additional subjects will be enrolled in an expansion cohort that will further evaluate ABT-700.
  Interventions: Drug: ABT-700
- Cohort B (Experimental): ABT-700 plus docetaxel.
  Interventions: Drug: ABT-700; Drug: docetaxel
- Cohort C (Experimental): ABT-700 plus FOLFIRI/cetuximab
  Interventions: Drug: ABT-700; Drug: FOLFIRI; Drug: cetuximab
- Cohort D (Experimental): ABT-700 plus erlotinib
  Interventions: Drug: ABT-700; Drug: erlotinib

INTERVENTIONS:
Drug: ABT-700 — ABT-700 will be administered by intravenous infusion at escalating dose levels on day 1 in 21-day dosing cycles. Additional subjects will be enrolled in an dose expansion cohort that will further evaluate ABT-700.
Drug: docetaxel — Docetaxel will be administered by intravenous infusion on Day 1 in 21-day dosing cycles.
  Arms: Cohort B
Drug: FOLFIRI — 5-fluorouracil, Folinic acid and Irinotecan will be administered by intravenous infusion on Day 1 and 15 in 28-day dosing cycles.
  Arms: Cohort C
Drug: cetuximab — Cetuximab will be administered by intravenous infusion weekly.
  Arms: Cohort C
Drug: erlotinib — Erlotinib will be taken orally daily.
  Arms: Cohort D
Drug: ABT-700 — ABT-700 will be administered by intravenous infusion on Day 1 and Day 15 in 28-day dosing cycles.
  Arms: Cohort C

SUMMARY:
This is a Phase 1/1b open-label study evaluating the safety, pharmacokinetics (PK), and preliminary efficacy of ABT-700 in subjects with advanced solid tumors that may have MET amplification or c-Met overexpression. ABT-700, previously known as h224G11 in publications, is an anti-c-Met antibody. The early clinical development plan for ABT-700 is based on the activity demonstrated in preclinical models. Up to 124 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subject with advanced solid tumors; Dose-expansion: evidence for MET gene amplification.
* Subject must have disease: a) that is not amenable to surgical resection, or b) that has progressed or recurred despite standard therapy, or c) that has failed to respond to standard therapy, or d) for which no effective therapy exists.
* Subject cannot tolerate or must not be eligible for other approved therapeutic options with known survival advantage.
* Subjects enrolled on the combination therapy phase must satisfy the above inclusion criteria and also the following: Subjects must have inoperable, locally advanced or metastatic cancer and be eligible to receive docetaxel or FOLFIRI/cetuximab or erlotinib in combination with ABT-700.

Exclusion Criteria:

* Subject has received anticancer therapy including chemotherapy, immunotherapy, radiation therapy, immunotherapy, biologic, or any investigational therapy within a period of 21 days, or herbal therapy within 7 days prior to the first dose of ABT-700.
* Subjects with uncontrolled metastases of the central nervous system. Subjects with brain metastases are eligible provided they have shown clinical and radiographic stable disease after definitive therapy and have not used steroids for at least 1 month prior to first dose of ABT-700.
* Subject has unresolved adverse events > Grade 1 from prior anticancer therapy except for alopecia or anemia.
* Subject has had major surgery within 21 days prior to the first dose of ABT-700.
* Subjects enrolled on the combination therapy phase must not meet the above exclusion criteria and must be eligible to receive docetaxel or FOLFIRI/cetuximab or erlotinib per most current prescribing information, or at the discretion of the Investigator. Subjects with K-Ras mutation-positive colorectal cancer will be excluded from receiving FOLFIRI/cetuximab.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-10-06 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ABT-700 when administered as monotherapy and in combination with docetaxel or 5-fluoruracil, folinic acid, irinotecan and cetuximab (FOLFIRI/cetuximab) or erlotinib | First cycle of treatment through 60 day follow-up visit
  Evaluation of vital signs, clinical lab testing, physical exams and adverse event monitoring
To Evaluate the pharmacokinetics of ABT-700 when administered as monotherapy and in combination with docetaxel or 5-fluoruracil, folinic acid, irinotecan and cetuximab (FOLFIRI/cetuximab) or erlotinib | At each cycle of treatment through 60 days after last dose.
  Pharmacokinetic profile of ABT-700 analyzed from blood samples
To determine the recommended Phase 2 dose for ABT-700 | First cycle of treatment through 60 day follow-up visit

SECONDARY OUTCOMES:
To evaluate the preliminary efficacy of ABT-700 when administered as monotherapy and in combination with docetaxel or 5-fluoruracil, folinic acid, irinotecan and cetuximab (FOLFIRI/cetuximab) or erlotinib | Screening through 60 day follow-up visit
  Objective response rate (complete and partial response), progression-free survival and duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Louie Naumovski, MD, Study Director — AbbVie